CLINICAL TRIAL: NCT07150520
Title: Acute Effects of Virtual Reality-Based Optokinetic Stimulation in Individuals With Multiple Sclerosis: Does Central Vestibular Dysfunction Alter These Effects?
Brief Title: VR-Based Optokinetic Stimulation in Multiple Sclerosis
Acronym: VR-OKS-MS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Avrasya University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özge Özdemir, M.Sc., Avrasya University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/102
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; vestibular dysfunction; optokinetic stimulation; virtual reality
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: All participants will receive the same virtual reality-based optokinetic stimulation protocol. Comparisons will be made between MS patients with and without central vestibular dysfunction and healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MS with Central Vestibular Dysfunction (Experimental): Participants with multiple sclerosis who have central vestibular dysfunction will receive a 10-minute session of virtual reality-based optokinetic stimulation (OKS) using Oculus Quest 2. Postural sway and motion sickness will be measured before and after the intervention.
  Interventions: Device: Virtual Reality-Based Optokinetic Stimulation (OKS)
- MS without Central Vestibular Dysfunction (Experimental): Participants with multiple sclerosis without central vestibular dysfunction will receive a 10-minute session of virtual reality-based optokinetic stimulation (OKS) using Oculus Quest 2. Postural sway and motion sickness will be measured before and after the intervention.
  Interventions: Device: Virtual Reality-Based Optokinetic Stimulation (OKS)
- Healthy Controls (Experimental): Healthy participants will receive a 10-minute session of virtual reality-based optokinetic stimulation (OKS) using Oculus Quest 2. Postural sway and motion sickness will be measured before and after the intervention
  Interventions: Device: Virtual Reality-Based Optokinetic Stimulation (OKS)

INTERVENTIONS:
Device: Virtual Reality-Based Optokinetic Stimulation (OKS) — A 10-minute session of virtual reality-based optokinetic stimulation (OKS) using the Oculus Quest 2 system. The stimulation speed is set at 40°/s and the direction is determined according to Fukuda test results. Postural sway and motion sickness will be assessed before and after the intervention.

SUMMARY:
The aim of this study is to investigate the acute effects of virtual reality-based optokinetic stimulation on postural sway and motion sickness symptoms in individuals with multiple sclerosis (MS)

DETAILED DESCRIPTION:
This study will be conducted at Hacettepe University, Faculty of Physical Therapy and Rehabilitation. It will investigate the acute effects of virtual reality-based optokinetic stimulation (OKS) on postural sway and motion sickness symptoms in individuals with multiple sclerosis (MS). Participants will include MS patients with and without central vestibular dysfunction, as well as age- and sex-matched healthy controls. MS participants will first undergo vestibular function assessment using videonystagmography (VNG). Postural control will then be measured via a force platform under four conditions (bipodal/monopodal, eyes open/closed) before and after a 10-minute OKS session using Oculus Quest 2. Healthy participants will follow the same postural and OKS assessment protocol without VNG.Motion sickness and virtual reality effects will be evaluated using the Simulator Sickness Questionnaire. Data will be analyzed using appropriate parametric or non-parametric tests to compare postural sway and VR-related symptoms across groups, with significance set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Be an adult aged 18-55 years
* Have a confirmed diagnosis of MS by a neurologist (for MS groups)
* Not have had a relapse in the last 3 months (for MS patients)
* Have an Expanded Disability Status Scale (EDSS) score of ≤ 4 (for MS patients)
* Be a healthy control with no condition preventing participation

Exclusion Criteria:

* Have peripheral vestibular dysfunction (for MS groups)
* Be older than 55 years
* Have any cardiovascular, orthopedic, neurological, or other condition preventing assessments
* Have a history of neurological disorders, head trauma, or chronic psychiatric conditions (for healthy controls)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Postural Sway | Immediately before and immediately after the 10-minute virtual reality-based optokinetic stimulation session
  Postural sway will be assessed using the FreeMED force platform under four conditions (bipodal/monopodal, eyes open/closed) before and after a 10-minute virtual reality-based optokinetic stimulation (OKS) session. Parameters include sway path, mediolateral (delta X), and anteroposterior (delta Y) displacement.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.meta.com/quest/